CLINICAL TRIAL: NCT03351010
Title: Thai Buddhism-based Mindfulness for Pain Management in Thai Outpatients With Cancer: A Pilot Study
Brief Title: Mindfulness for Pain Management in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Srisuda Ngamkham, Nursing Instructor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12/2561
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Cancer, Metastatic; Pain, Chronic
Keywords: Mindfulness, Cancer, Pain Management
MeSH Terms: conditions — Neoplasm Metastasis; Chronic Pain; Neoplasms; Agnosia

STUDY DESIGN:
Intervention Model Description: Using a randomized controlled trial design, the investigators will test theTBbM intervention to improve pain in Thai outpatients (N=160) with cancer who are receiving cancer care at Sawanpracharak Hospital, Thailand. The control group (n = 80) will receive usual care and participate in a one-hour video educational program about cancer pain. The intervention group (n = 80) will receive usual care, participate in a one-hour video educational program about cancer pain, and receive an 8-week TBbM intervention.
Who Masked: Participant
Masking Description: Eligible patients will 1) have any cancer type or stage, 2) be 18-60 years of age, 3) have a worst pain score > 4 in the past 7 days, 4) be able to read and write the Thai language, 5) have a Karnofsky Performance status > 70%, and be willing to travel to the temple. Exclusion criteria will be any diagnosed psychiatric illness that would prevent the patient from giving informed consent or from participating fully in the study. Patients with comorbidities (e.g., arthritis, bone metastasis, deformity, certain neurologic conditions such as biracial plexus nerve compression) that would impair the ability to perform the hand and arm movements also are ineligible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Receiving education program and mindfulness training
  Interventions: Behavioral: Mindfulness training program; Device: Cancer pain educational program
- Control (Active Comparator): Receiving education program
  Interventions: Device: Cancer pain educational program

INTERVENTIONS:
Behavioral: Mindfulness training program — The mindfulness training program is a self-awareness mindfulness training program by performing the 15-position hand movement series
  Arms: Mindfulness
Device: Cancer pain educational program — A cancer pain education program by using Videos and personalized face-to-face techniques

SUMMARY:
Using pharmacologic agents are often effective to treat patients with cancer pain, but there are associated with serious side-effects and risks of dependence and addiction. The Thai Buddhism-based Mindfulness (TBbM) intervention created by a widely respected Buddhist monk focuses on testing a meditation technique to manage pain. If effective, millions of patients who suffer with cancer pain will benefit from use of a safe, culturally appropriate, non-pharmacologic approach to pain management.

DETAILED DESCRIPTION:
Cancer is leading cause of death in Thailand. One hundred and twenty-eight men and 83 women per 100,000 had a common consequence both of malignancy and its treatment. Pain is experienced by 62% of Thai patients with cancer. Cancer pain is a major health problem because it causes both physical and psychological suffering for millions of individuals. Although pharmacological/analgesic treatment is effective, adverse side effects are common. Internationally, mindfulness is being used as an effective non-pharmacological treatment for psychological problems including distress, anxiety, stress, depression, and to improve quality of life in patients with cancer. However, the effect of mindfulness on pain as the primary outcome has not been sufficiently investigated. A few randomized controlled trials provide evidence that mindfulness interventions influence pain intensity in patients with cancer pain, but culturally targeted interventions have not been tested. Therefore, the purpose of this research is to test the effect of the Thai Buddhism-based Mindfulness (TBbM) program for pain management in Thai outpatients. Using a randomized controlled trial design, the investigators will test theTBbM intervention to improve pain in Thai outpatients (N=160) with cancer who are receiving cancer care at Sawanpracharak Hospital, Thailand. The control group (n = 80) will receive usual care and participate in a one-hour video educational program about cancer pain. The intervention group (n = 80) will receive usual care, participate in a one-hour video educational program about cancer pain, and receive an 8-week TBbM intervention. Investigators will accomplish the overall objective by pursuing the following three specific aims: 1) to compare the effect of the TBbM intervention to that of usual care on worst pain severity (primary outcome) as measured by the Brief Pain Inventory Thai Version (BPI-T); 2) to compare the effect of the TBbM intervention to that of usual care on secondary outcomes (i.e., pain interference, average pain, anxiety and depression, mindfulness, locus of control, and QoL) as measured by the BPI-T, the Hospital Anxiety and Depression Scale Thai Version (HADS-T), the Mindfulness Assessment Scale Thai Version (MAS-T), the Beliefs in Pain Control Questionnaire Thai Version (BPCQ-T) and the Functional Assessment of Cancer Therapy-General-Thai Version (FACT-G-T); and 3) to explore the mediating effects of TBbM-induced changes in cognitive (locus of control) and psychological factors (anxiety and depression) on worst pain severity. The investigators posit that the TBbM intervention will be more effective than usual care in reducing pain (primary outcome) and improving pain interference, anxiety, depression, mindfulness, locus of control, and QoL (secondary outcomes). T-tests, analysis of covariance (ANOVA), and path analysis approaches will be used to evaluate TBbM outcomes.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will:

* have any cancer type or stage,
* be 18-60 years of age,
* have a worst pain score > 4 in the past 7 days,
* be able to read and write the Thai language,
* have a Karnofsky Performance status > 70%, and
* be willing to travel to the temple.

Exclusion Criteria:

* Patients will be diagnosed psychiatric illness
* Patients will have the comorbidities (e.g., arthritis, bone metastasis, deformity, certain neurological conditions such as Brachial plexus nerve compression)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Pain Change Over Time | Baseline, 4 weeks and 8 weeks
  Worst pain scores are measured by Brief Pain Inventory. The Brief Pain Inventory-Short Form asks about pain in general, pain location, pain intensity (worst, least, average, and present), and is scored on a numerical rating scale of 0 (no pain) to 10 (pain as bad as one can imagine.

SECONDARY OUTCOMES:
Pain | Baseline and 8 weeks
  Pain interference and average pain scores are measured by the Brief Pain Inventory
Anxiety and depression | Baseline and 8 weeks
  Anxiety and depression scores are measured by the Hospital Anxiety and Depression Scale
Mindfulness | Baseline and 8 weeks
  Mindfulness scores are measured by the Mindfulness Assessment Scale
Locus of control | Baseline and 8 weeks
  Personal control scores are measured by the Beliefs in Pain Control Questionnaire
Quality of life | Baseline and 8 weeks
  Quality of life scores are measured by the Functional Assessment of Cancer Therapy-General-Thai Version

CONTACTS AND LOCATIONS:
Locations (1):
- Sawanpracharak Hospital, Maung, Nakhonsawan, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The individual data of the participants that we will collect are cancer data, treatment data, and a time period of mindfulness practice
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 8 weeks
Access Criteria: Eligible patients will 1) have any cancer type or stage, 2) be 18-60 years of age, 3) have a worst pain score > 4 in the past 7 days, 4) be able to read and write the Thai language, 5) have a Karnofsky Performance status > 70%, and be willing to travel to the temple.
URL: http://www.umich.edu

REFERENCES:
- [Result] Fish JA, Ettridge K, Sharplin GR, Hancock B, Knott VE. Mindfulness-based cancer stress management: impact of a mindfulness-based programme on psychological distress and quality of life. Eur J Cancer Care (Engl). 2014 May;23(3):413-21. doi: 10.1111/ecc.12136. Epub 2013 Oct 10. PMID 24118428